CLINICAL TRIAL: NCT01128985
Title: A Double-Blind, Placebo-Controlled, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Multiple Dose Pharmacokinetic and Pharmacodynamic Characteristics of JNJ-28431754 (Canagliflozin) in Subjects With Type 2 Diabetes Mellitus
Brief Title: A Pharmacokinetic and Pharmacodynamic Study to Determine Blood Levels of JNJ-28431754 (Canagliflozin) in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR017200; 28431754DIA1023
Record Dates: First submitted 2010-05-20; First posted 2010-05-24 (Estimated); Last update posted 2013-05-29 (Estimated); Status verified 2013-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Canagliflozin; Placebo; Type 2 diabetes mellitus; Pharmacokinetic; Pharmacodynamic
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Canagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (4):
- 001 (Experimental): Canagliflozin 50 mg 50 mg capsule once daily for 7 consecutive days from Day 1 to Day 7
  Interventions: Drug: Canagliflozin 50 mg
- 002 (Experimental): Canagliflozin 100 mg 100 mg capsule once daily for 7 consecutive days from Day 1 to Day 7
  Interventions: Drug: Canagliflozin 100 mg
- 003 (Experimental): Canagliflozin 300 mg 300 mg capsule once daily for 7 consecutive days from Day 1 to Day 7.
  Interventions: Drug: Canagliflozin 300 mg
- 004 (Placebo Comparator): Placebo matching canagliflozin placebo once daily for 7 consecutive days from Day 1 to Day 7
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Canagliflozin 50 mg — 50 mg capsule once daily for 7 consecutive days from Day 1 to Day 7
  Arms: 001
Drug: Canagliflozin 100 mg — 100 mg capsule once daily for 7 consecutive days from Day 1 to Day 7
  Arms: 002
Drug: Canagliflozin 300 mg — 300 mg capsule once daily for 7 consecutive days from Day 1 to Day 7.
  Arms: 003
Drug: Placebo — matching canagliflozin placebo once daily for 7 consecutive days from Day 1 to Day 7
  Arms: 004

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (blood levels of the drug) and pharmacodynamics (effects of the drug on the body) of canagliflozin after oral administration to patients with type 2 diabetes mellitus.

DETAILED DESCRIPTION:
Canagliflozin is a drug that is being tested to see if it may be useful in treating patients diagnosed with type 2 diabetes mellitus (T2DM). This is a randomized (patients will assigned to 1 of 4 study treatments by chance), double-blind (neither the patient or the study doctor will know the name of the assigned treatment), study to assess the pharmacokinetics (blood levels) and pharmacodynamics (effects of the drug on the body) of canagliflozin compared to a placebo (a capsule that looks like all the other treatments but has no real medicine) in patients with T2DM. Approximately 36 patients with T2DM will receive once-daily treatment with canagliflozin (50 mg, 100 mg, or 300 mg doses) or placebo for 7 days. Patients will participate in the study for approximately 9 weeks. Blood and urine samples will be collected at specified times before and after each dose of study drug for pharmacokinetic and pharmacodynamic analyses. A blood sample will also be collected before the first dose of study drug for pharmacogenomic analysis (ie, genetic testing) for possible use in characterizing the safety and/or efficacy of study drug in relation to the patient pharmacogenic profile. During the study, the safety and tolerability of canagliflozin will be evaluated by monitoring adverse events and findings from laboratory evaluations, vital signs measurements, and ECG measurements. The primary outcome measure in the study is the concentration of canagliflozin and its major metabolites (M5 and M7) in the blood measured by protocol-specified pharmacokinetic parameters at protocol specified time points through Day 7. Study drug will be taken orally (by mouth) once daily before the first meal each day. On Day -1, patients will take 1 dose of placebo in single-blind fashion (patient blinded) to determine baseline assessments. After randomization, patients will take single doses of double-blind canagliflozin (50 mg, 100 mg, or 300 mg) or matching placebo once daily for 7 days (Day 1 through Day 7).

ELIGIBILITY:
Inclusion Criteria:

* All patients must have a diagnosis of T2DM for at least 1 year, but not more than 12 years prior to Day -1 of the study and be medically stable on the basis of physical examination, medical history, laboratory safety test results, vital signs and electrocardiogram (ECG) performed at Screening
* Patients must be on generally stable approved anti-hypeglycemic agent (AHA) regimen (i.e., with no change in medication, or only 1 dose step change in dose) for at least 2 months prior to the Screening Visit
* Patients must have fasting plasma glucose (FPG) concentrations between 7.8 mM (140 mg/dL) and 15 mM (270 mg/dL) on Day -2

Exclusion Criteria:

* History of clinically significant diabetic complications including retinopathy, nephropathy, or macro albuminuria, neuropathy, gastroparesis, or diabetic ketoacidosis
* History of type 1 diabetes mellitus (T1DM)
* History of repeated severe hypoglycemic episodes before screening

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-03; Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
The concentration of canagliflozin and major metabolites (M5 and M7) in blood will be measured by protocol-specified pharmacokinetic parameters. | At protocol-specified time points through Day 7

SECONDARY OUTCOMES:
The relationship between the concentration of glucose in patient blood measured by protocol-specified pharmacodynamic parameters | At protocol-specified time points from baseline to Day 7
The safety and tolerability of canagliflozin will be determined by monitoring adverse events and findings from laboratory evaluations, vital signs measurements, and ECG measurements reported. | At protocol-specified time points from the time of screening (Day -44 to Day -23) to end-of-study (7 to 10 days after Day 7 or at the time of early withdrawal from the study)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.
Locations (2):
- United States (2):
  - Fort Myers, Florida
  - Miramar, Florida

REFERENCES:
- See also: A Double-blind, Placebo-Controlled, Randomized, Parallel-Group, Multi-Center Study to Evaluate the Multiple-Dose Pharmacokinetic and Pharmacodynamic Characteristics of JNJ-28431754 (Canagliflozin) in Subjects With Type 2 Diabetes Mellitus — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=857&filename=CR017200_CSR.pdf